CLINICAL TRIAL: NCT06628479
Title: Relaxin, Matrix Metalloproteinase-2 and Interleukin-6 in Women With Chronic Pelvic Pain, Diagnosis of Deep Infiltrative Endometriosis and Investigation of it is Place in Follow-up
Brief Title: Relaxin, Matrix Metalloproteinase-2 and Interleukin-6 in Women With Chronic Pelvic Pain
Status: Completed | Type: Observational
Sponsor: Sanliurfa Mehmet Akif Inan Education and Research Hospital (Other)
Collaborators: University of Health Sciences School of Medicine Bursa Yuksek Ihtisas Research and Training Hospital, Department of Obstetrics and Gynecology, Bursa, Turkey (Unknown)
Responsible Party: Principal Investigator, Nefise Nazlı YENIGUL, Ph.D. Assistant Professor Department of Obstetrics and Gynecology, Sanliurfa Mehmet Akif Inan Education and Research Hospital
Other Study IDs: 2011-KAEK-25 2022/05-18
Record Dates: First submitted 2024-06-09; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Endometriosis
Keywords: Chronic pelvic pain; Deep infiltrative endometriosis; Relaxin; IL-6; MMP-2
MeSH Terms: conditions — Endometriosis | interventions — Interleukins; Enzymes; Hormones; Relaxin; Matrix Metalloproteinase 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Deep infiltrative endometriosis group: People over the age of 35 who have completed their fertility, do not want children and have chronic pelvic endometriosis with pain or patients diagnosed with adenomyosis due to abnormal uterine bleeding
  Interventions: Other: interleukin, enzyme, hormone
- control group: Patients operated for tubal ligation without pelvic pain
  Interventions: Other: interleukin, enzyme, hormone

INTERVENTIONS:
Other: interleukin, enzyme, hormone — Relaxin, MMP-2 and IL-6 values from vaginal washing fluid, peritoneal washing fluid and serum samples
  Other Names: relaxin; mmp-2; ıl-6

SUMMARY:
In our study, by evaluating the serum and vaginal-peritoneal fluid levels of Relaxin, Matrix Metalloproteinase-2 and Interleukin-6 in women over 35 years of age with chronic pelvic pain, the investigators aimed to reveal their potential to be an important marker in the diagnosis of Deep Infiltrative Endometriosis, thus enabling early diagnosis with lower cost and results that can be obtained in a short time.The investigators aim to reveal its relationship with follow-up.

In our study, the values of Relaxin, MMP-2 or IL-6 from vaginal fluids were found to be significantly higher than the control group in the prediction and follow-up of deep infiltrative endometriosis. This supports the role of Relaxin and MMP-2 as well as IL-6 in the pathophysiology of deep infiltrative endometriosis.

Histologically based and multicenter randomized controlled studies with more patients are needed to elucidate the etiology and pathophysiology of endometriosis.

DETAILED DESCRIPTION:
10 cc of vaginal washing fluid, serum samples on the day of operation and 20 cc of pelvic washing fluid during laparoscopy were taken from all patients before the operation. Patients were included in the FA group according to the ENZIAN Classification. Patients' age, BMI, gravida, parity, obstetric history such as pregnancy, ethnic origin, educational status, preoperative and postoperative evaluation for chronic pelvic pain, laboratory tests (routine tests such as Ca125, CRP, FSH, LH, E2, P), Preoperative and postoperative hormonal values were recorded. Relaxin, MMP-2 and IL-6 values from vaginal washing fluid, peritoneal washing fluid and serum samples of the patients in the control and study groups were compared.

ELIGIBILITY:
Inclusion Criteria:

Endometriosis patients Adenomyosis patients

Exclusion Criteria:

Ovarian endometriosis Chronic pelvic pain with another reason

Ages: 35 Years to 72 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People over the age of 35 who have completed their fertility, do not want children and have chronic pelvic patients with pain
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Investigation of the role of Relaxin, Matrix Metalloproteinase-2 and Interleukin 6 in the diagnosis and follow-up of deep infiltrative endometriosis in women with chronic pelvic pain | 6 months
  Quantitative levels of Relaxin, MMP-2, and IL-6 in serum will be measured. The levels of these biomarkers will be reported as concentrations in nanograms per milliliter (ng/mL) for serum. These measurements aim to establish the correlation between biomarker levels and the presence of Deep Infiltrative Endometriosis (DIE) in women over 35 years of age with chronic pelvic pain.
Investigation of the role of Relaxin, Matrix Metalloproteinase-2 and Interleukin 6 in the diagnosis and follow-up of deep infiltrative endometriosis in women with chronic pelvic pain | 6 months
  Quantitative levels of Relaxin, MMP-2, and IL-6 in vaginal-peritoneal fluid will be measured. The levels of these biomarkers will be reported as concentrations in micromoles per liter (µmol/L) for vaginal-peritoneal fluid. These measurements aim to establish the correlation between biomarker levels and the presence of Deep Infiltrative Endometriosis (DIE) in women over 35 years of age with chronic pelvic pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Nefise Nazlı YENIGUL, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No